CLINICAL TRIAL: NCT03730909
Title: The Effect of Lactate Administration on Cerebral Blood Flow During Hypoglycemia; Are the Suppressive Effects of Lactate on Counterregulatory Responses to Hypoglycemia Reflected in an Altered CBF Response?
Brief Title: The Effect Lactate Administration on Cerebral Blood Flow During Hypoglycemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Lactate_CBF
Record Dates: First submitted 2018-10-22; First posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-10

CONDITIONS: Type1diabetes; Hypoglycemia Unawareness
MeSH Terms: interventions — Sodium Lactate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactate infusion (Experimental): Subjects will receive an intravenous lactate infusion to elevate plasma lactate levels
  Interventions: Drug: Sodium Lactate
- NaCl infusion (Placebo Comparator): As a control condition, subjects will receive intravenous NaCl infusion
  Interventions: Drug: Sodium chloride

INTERVENTIONS:
Drug: Sodium Lactate — IV infusion
  Arms: Lactate infusion
Drug: Sodium chloride — IV infusion
  Arms: NaCl infusion

SUMMARY:
It is thought that altered brain lactate handling is involved in the development of impaired awareness of hypoglycemia (IAH), i.e. the inability to timely detect hypoglycemia in people with type 1 diabetes (T1DM). Infusion of lactate diminishes symptomatic and hormonal responses to hypoglycemia in patients with normal awareness of hypoglycemia (NAH), resembling the situation of patients with IAH. It is unknown whether this attenuating effect is due to brain lactate oxidation or the result of lactate-induced alterations of global and regional cerebral blood flow (CBF).

Normally, hypoglycemia causes a redistribution of CBF towards the thalamus, from where the sympathetic response to hypoglycemia is coordinated, but in IAH this effect is absent and global CBF is increased. We hypothesize that lactate infusion in patients with NAH will result in blunting of thalamic activation and/or enhanced global CBF. If so, these results may help delineating the pathogenesis of IAH which eventually creates new avenues to protect against the morbidity associated with hypoglycemia and IAH.

Study design: Single-blind placebo controlled, randomized cross-over intervention study Study population: T1DM patients with NAH (n=10) Intervention: On two separate occasions, patients with T1DM and NAH will undergo a hyperinsulinemic euglycemic-hypoglycemic glucose clamp with or without the infusion of exogenous lactate. ASL-MRI will be applied to measure global and regional changes in CBF.

Main study parameters/endpoints: The change in regional thalamic CBF in response to intravenous lactate infusion compared to placebo, during hypoglycemia

ELIGIBILITY:
Inclusion Criteria:

* Diabetes duration ≥ 1 year
* Age: 18-50 years
* Body-Mass Index: 18-30 kg/m2
* HbA1c: 42-75 mmol/mol (6-9%)
* Outcome Clarke questionnaire: 0-1
* Blood pressure: <160/90 mmHg

Exclusion Criteria:

* Inability to provide informed consent
* Use medication other than insulin, except for oral contraceptives or stable thyroxin supplementation therapy
* Presence of any other medical condition that might interfere with the study protocol, such as brain injuries, epilepsy, a major cardiovascular disease event or cardiac failure, known liver disease, anxiety disorders or a history of panic attacks.
* Microvascular complications of T1DM: Proliferative retinopathy, symptomatic diabetic neuropathy (including autonomic neuropathy) or Nephropathy; clinical/overt albuminuria or an estimated glomerular filtration rate <60ml/min/1.73m2.
* MRI contraindications (pregnancy, severe claustrophobia, metal parts in body)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-06-11 (Actual); Primary Completion 2019-04-11 (Estimated); Study Completion 2019-06-11 (Estimated)

PRIMARY OUTCOMES:
Regional CBF in ml/100g/min measured with ASL-MRI | during stable euglycemia (40 minutes) and hypoglycemia (45 minutes)
  The change in regional thalamic CBF in response to intravenous lactate infusion compared to placebo, during hypoglycemia

SECONDARY OUTCOMES:
Global CBF in ml/100g/min measured with ASL-MRI | during stable euglycemia (40 minutes) and hypoglycemia (45 minutes)
  The change in global CBF in response to intravenous lactate infusion
Counterregulatory hormone responses to hypoglycemia | during stable euglycemia (40 minutes) and hypoglycemia (45 minutes)
  The difference in adrenaline (pmol/L) responses to hypoglycemia during lactate infusion compared to placebo
Symptom responses to hypoglycemia | during stable euglycemia (40 minutes) and hypoglycemia (45 minutes)
  The difference in symptom responses to hypoglycemia (meausured with a validated questionnaire) during lactate infusion compared to placebo
Measurements of metabolites in cell lysates or supernatants of the cultured immune cells | during stable euglycemia (40 minutes) and hypoglycemia (45 minutes)
  The effect of lactate administration on immune cell function and metabolism

CONTACTS AND LOCATIONS:
Locations (1):
- Radoud university medical center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van Meijel LA, van Asten JJA, Grandjean J, Heerschap A, Tack CJ, van der Graaf M, Wiegers EC, de Galan BE. Effect of lactate administration on cerebral blood flow during hypoglycemia in people with type 1 diabetes. BMJ Open Diabetes Res Care. 2022 Mar;10(2):e002401. doi: 10.1136/bmjdrc-2021-002401. PMID 35321886